CLINICAL TRIAL: NCT06051526
Title: The African Critical Illness Outcomes Study
Acronym: ACIOS
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Co-chief Investigator, University of Cape Town
Other Study IDs: ACIOS
Record Dates: First submitted 2023-09-01; First posted 2023-09-25 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness; Mortality
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill in-patients: All adult inpatients in hospitals across Africa that are critically ill.

SUMMARY:
In Africa, the prevalence of critical illness is likely to be higher due to a greater burden of disease, and the associated mortality higher due to limited resources. This is a prospective, observational study to rapidly establish the prevalence of critical illness in in-hospital adult patients in Africa, and the resources available to provide essential critical care (care that should be available to every patient in the world) and factors associated with mortality. Rapid dissemination of these findings may help mitigate mortality from critical illness in Africa. These points provide the rationale for the African Critical Illness Outcomes Study.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

The objectives of this study are to determine:

1. The proportion of hospital patients who are critically ill,
2. The mortality associated with critical illness,
3. The proportion of critically ill patients who receive essential emergency and critical care,
4. The relationship between essential emergency and critical care provision, and mortality, and
5. The availability of resources necessary to provide essential emergency and critical care.

STUDY DESIGN

An African multi-centre prospective observational cohort study of adult (≥18 years) in-hospital patients. Patient follow up will be for a maximum of 7 days in-hospital.

The primary outcome is in-hospital mortality in adult hospital patients with and without critical illness in Africa.

The intention is to provide a representative sample of the mortality, the risk factors associated with mortality in adult patients with critical illness, and the resources available and interventions provided to treat critical illness in Africa. This study will run between September and November 2023.

PREPARATORY WORK

This study will be run by the African Perioperative Research Group (APORG), with a network of over 600 hospitals in more than 40 African countries which has successfully conducted the African Surgical Outcomes Study (ASOS), the ASOS-2 Trial, the African COVID-19 Critical Care Outcomes Study (ACCCOS) and the African Pediatric Surgical Outcomes Study (ASOS-PEDS).

IMPORTANCE OF THIS STUDY

To decrease the mortality associated with critical illness in Africa, it is important to rapidly establish the potential risk factors for mortality, and resources available to manage these patients. The APORG network has the capacity to provide these data timeously.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 years or over who have been admitted for inpatient care in any department or ward in participating hospitals.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients aged 18 years or over who have been admitted for inpatient care in any department or ward in participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 20159 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Presence of critical illness | 7 days
  The number of participants with critical illness.
In-hospital mortality (censored at 7-days) | 7 days
  The number of participants with in-hospital mortality (censored at 7-days)

SECONDARY OUTCOMES:
Provision of essential emergency and critical care | 7 days
  To number of critically ill patients who receive essential emergency and critical care.
Length of hospital stay | 7 days
  The length of hospital stay for critically ill patients
Number of essential emergency and critical care resources available for care | 7 days
  The number of essential emergency and critical care resources available

CONTACTS AND LOCATIONS:
Overall Officials: Tim Baker, MBChB; PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Merowe Daman Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes
A pragmatic and realistic dataset is fundamental to the success of the study. Data will be collected on paper on one-day in each hospital plus follow-up censored at 7 day.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from the time of publication and for 10 years following publication.
Access Criteria: Contributing researchers and collaborators
URL: https://www.asos.org.za/index.php/acios

REFERENCES:
- [Result] Kayambankadzanja RK, Schell CO, Gerdin Warnberg M, Tamras T, Mollazadegan H, Holmberg M, Alvesson HM, Baker T. Towards definitions of critical illness and critical care using concept analysis. BMJ Open. 2022 Sep 5;12(9):e060972. doi: 10.1136/bmjopen-2022-060972. PMID 36606666
- [Result] Jenson A, Hansoti B, Rothman R, de Ramirez SS, Lobner K, Wallis L. Reliability and validity of emergency department triage tools in low- and middle-income countries: a systematic review. Eur J Emerg Med. 2018 Jun;25(3):154-160. doi: 10.1097/MEJ.0000000000000445. PMID 28263204
- [Result] Kruisselbrink R, Kwizera A, Crowther M, Fox-Robichaud A, O'Shea T, Nakibuuka J, Ssinabulya I, Nalyazi J, Bonner A, Devji T, Wong J, Cook D. Modified Early Warning Score (MEWS) Identifies Critical Illness among Ward Patients in a Resource Restricted Setting in Kampala, Uganda: A Prospective Observational Study. PLoS One. 2016 Mar 17;11(3):e0151408. doi: 10.1371/journal.pone.0151408. eCollection 2016. PMID 26986466
- [Result] Phua J, Faruq MO, Kulkarni AP, Redjeki IS, Detleuxay K, Mendsaikhan N, Sann KK, Shrestha BR, Hashmi M, Palo JEM, Haniffa R, Wang C, Hashemian SMR, Konkayev A, Mat Nor MB, Patjanasoontorn B, Nafees KMK, Ling L, Nishimura M, Al Bahrani MJ, Arabi YM, Lim CM, Fang WF; Asian Analysis of Bed Capacity in Critical Care (ABC) Study Investigators, and the Asian Critical Care Clinical Trials Group. Critical Care Bed Capacity in Asian Countries and Regions. Crit Care Med. 2020 May;48(5):654-662. doi: 10.1097/CCM.0000000000004222. PMID 31923030
- [Result] Maharaj R, Raffaele I, Wendon J. Rapid response systems: a systematic review and meta-analysis. Crit Care. 2015 Jun 12;19(1):254. doi: 10.1186/s13054-015-0973-y. PMID 26070457
- [Result] Kayambankadzanja RK, Likaka A, Mndolo SK, Chatsika GM, Umar E, Baker T. Emergency and critical care services in Malawi: Findings from a nationwide survey of health facilities. Malawi Med J. 2020 Mar;32(1):19-23. doi: 10.4314/mmj.v32i1.5. PMID 32733655
- [Result] Baker T, Lugazia E, Eriksen J, Mwafongo V, Irestedt L, Konrad D. Emergency and critical care services in Tanzania: a survey of ten hospitals. BMC Health Serv Res. 2013 Apr 16;13:140. doi: 10.1186/1472-6963-13-140. PMID 23590288
- [Result] Kayambankadzanja RK, Schell CO, Mbingwani I, Mndolo SK, Castegren M, Baker T. Unmet need of essential treatments for critical illness in Malawi. PLoS One. 2021 Sep 10;16(9):e0256361. doi: 10.1371/journal.pone.0256361. eCollection 2021. PMID 34506504
- [Result] Schell CO, Gerdin Warnberg M, Hvarfner A, Hoog A, Baker U, Castegren M, Baker T. The global need for essential emergency and critical care. Crit Care. 2018 Oct 29;22(1):284. doi: 10.1186/s13054-018-2219-2. PMID 30373648
- [Result] Crawford AM, Shiferaw AA, Ntambwe P, Milan AO, Khalid K, Rubio R, Nizeyimana F, Ariza F, Mohammed AD, Baker T, Banguti PR, Madzimbamuto F. Global critical care: a call to action. Crit Care. 2023 Jan 20;27(1):28. doi: 10.1186/s13054-022-04296-3. PMID 36670506
- [Result] Mekontso Dessap A, Richard JM, Baker T, Godard A, Carteaux G. Technical Innovation in Critical Care in a World of Constraints: Lessons from the COVID-19 Pandemic. Am J Respir Crit Care Med. 2023 May 1;207(9):1126-1133. doi: 10.1164/rccm.202211-2174CP. PMID 36716353
- [Result] Buowari DY, Owoo C, Gupta L, Schell CO, Baker T; EECC Network Group. Essential Emergency and Critical Care: A Priority for Health Systems Globally. Crit Care Clin. 2022 Oct;38(4):639-656. doi: 10.1016/j.ccc.2022.06.008. PMID 36162903
- [Result] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Result] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Result] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Lancet. 2015 Aug 8;386(9993):569-624. doi: 10.1016/S0140-6736(15)60160-X. Epub 2015 Apr 26. No abstract available. PMID 25924834
- [Result] Murthy S, Wunsch H. Clinical review: International comparisons in critical care - lessons learned. Crit Care. 2012 Dec 12;16(2):218. doi: 10.1186/cc11140. PMID 22546146
- [Result] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Result] African COVID-19 Critical Care Outcomes Study (ACCCOS) Investigators. Patient care and clinical outcomes for patients with COVID-19 infection admitted to African high-care or intensive care units (ACCCOS): a multicentre, prospective, observational cohort study. Lancet. 2021 May 22;397(10288):1885-1894. doi: 10.1016/S0140-6736(21)00441-4. PMID 34022988
- [Result] Ilori IU, Kalu QN. Intensive care admissions and outcome at the University of Calabar Teaching Hospital, Nigeria. J Crit Care. 2012 Feb;27(1):105.e1-4. doi: 10.1016/j.jcrc.2011.11.011. PMID 22304993
- [Result] Towey RM, Ojara S. Practice of intensive care in rural Africa: an assessment of data from Northern Uganda. Afr Health Sci. 2008 Mar;8(1):61-4. No abstract available. PMID 19357737
- [Result] Gombar S, Ahuja V, Jafra A. A retrospective analysis of obstetric patient's outcome in intensive care unit of a tertiary care center. J Anaesthesiol Clin Pharmacol. 2014 Oct;30(4):502-7. doi: 10.4103/0970-9185.142843. PMID 25425775
- [Result] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Result] Kause J, Smith G, Prytherch D, Parr M, Flabouris A, Hillman K; Intensive Care Society (UK); Australian and New Zealand Intensive Care Society Clinical Trials Group. A comparison of antecedents to cardiac arrests, deaths and emergency intensive care admissions in Australia and New Zealand, and the United Kingdom--the ACADEMIA study. Resuscitation. 2004 Sep;62(3):275-82. doi: 10.1016/j.resuscitation.2004.05.016. PMID 15325446
- [Result] Smith AF, Wood J. Can some in-hospital cardio-respiratory arrests be prevented? A prospective survey. Resuscitation. 1998 Jun;37(3):133-7. doi: 10.1016/s0300-9572(98)00056-2. PMID 9715771
- [Result] Kellett J, Deane B. The Simple Clinical Score predicts mortality for 30 days after admission to an acute medical unit. QJM. 2006 Nov;99(11):771-81. doi: 10.1093/qjmed/hcl112. Epub 2006 Oct 17. PMID 17046859
- [Result] Baker T, Blixt J, Lugazia E, Schell CO, Mulungu M, Milton A, Castegren M, Eriksen J, Konrad D. Single Deranged Physiologic Parameters Are Associated With Mortality in a Low-Income Country. Crit Care Med. 2015 Oct;43(10):2171-9. doi: 10.1097/CCM.0000000000001194. PMID 26154933
- [Result] Baker T, Gerdin M. The clinical usefulness of prognostic prediction models in critical illness. Eur J Intern Med. 2017 Nov;45:37-40. doi: 10.1016/j.ejim.2017.09.012. Epub 2017 Sep 19. PMID 28935477
- [Result] International Surgical Outcomes Study group. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. Br J Anaesth. 2016 Oct 31;117(5):601-609. doi: 10.1093/bja/aew316. PMID 27799174
- [Result] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Result] Baker T, Schell CO, Lugazia E, Blixt J, Mulungu M, Castegren M, Eriksen J, Konrad D. Vital Signs Directed Therapy: Improving Care in an Intensive Care Unit in a Low-Income Country. PLoS One. 2015 Dec 22;10(12):e0144801. doi: 10.1371/journal.pone.0144801. eCollection 2015. PMID 26693728
- [Result] Bell MB, Konrad D, Granath F, Ekbom A, Martling CR. Prevalence and sensitivity of MET-criteria in a Scandinavian University Hospital. Resuscitation. 2006 Jul;70(1):66-73. doi: 10.1016/j.resuscitation.2005.11.011. Epub 2006 Jun 6. PMID 16757089
- [Result] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- [Result] ASOS-2 Investigators. Enhanced postoperative surveillance versus standard of care to reduce mortality among adult surgical patients in Africa (ASOS-2): a cluster-randomised controlled trial. Lancet Glob Health. 2021 Oct;9(10):e1391-e1401. doi: 10.1016/S2214-109X(21)00291-6. Epub 2021 Aug 19. PMID 34418380

DOCUMENTS (3):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT06051526/Prot_000.pdf
  • Statistical Analysis Plan: Main study statistical analysis plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT06051526/SAP_001.pdf
  • Statistical Analysis Plan: Pain substudy statistical analysis plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT06051526/SAP_002.pdf